CLINICAL TRIAL: NCT02867436
Title: The Effect of Gluten-free Diet on Residual Beta-cell Capacity, Immune Function and Gut Microbiome in Children With Newly Diagnosed Type 1 Diabetes (T1D)
Brief Title: The Effect of Gluten-free Diet on New Onset Type 1 Diabetes (T1D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Zdeněk Šumník, MD, PhD, University Hospital, Motol
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-27994A
Record Dates: First submitted 2016-03-07; First posted 2016-08-16 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten-free diet (Experimental): Gluten-free diet
  Interventions: Other: Gluten-free diet
- Conventional diet (No Intervention): Conventional diet

INTERVENTIONS:
Other: Gluten-free diet
  Arms: Gluten-free diet

SUMMARY:
The primary aim of this pilot study is to test whether gluten-free diet (GFD) instituted in children shortly after onset of Type 1 Diabetes (T1D) can decelerate the decline in beta cell function as compared to age matched controls. Primary objective of the trial is the change in C-peptide area under the curve measured by mixed-meal tolerance test (MMTT) between group on GFD and standard gluten-containing diet.

Secondary objectives are:

* Changes in immune parameters between gluten-free diet group and control group;
* Differences in fecal microbiome between children on normal diet and children on GFD;

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes (T1D) diagnosed according to the American Diabetes Association criteria

Exclusion Criteria:

* negativity of the three diabetes-related autoantibodies at T1D onset;
* negativity of celiac-disease high risk Human Leucocyte Antigen DQB1 (HLA-DQB1) and Human Leucocyte Antigen DQA1 (HLA-DQA1) genotype HLA-DQB1*03:02-DQA1*03 nor DQB1*02-DQA1*05 molecules;
* celiac disease or positive transglutaminase antibody test;
* body mass index over two standard deviations of the age and height standard;
* any concomitant disease potentially influencing immune response or gluten sensitivity

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - University Hospital Královské Vinohrady, Prague
  - University Hospital Motol, Prague

REFERENCES:
- [Derived] Neuman V, Pruhova S, Kulich M, Kolouskova S, Vosahlo J, Romanova M, Petruzelkova L, Havlik J, Mascellani A, Henke S, Sumnik Z, Cinek O. Changes in the gut bacteriome upon gluten-free diet intervention do not mediate beta cell preservation. Diabetologia. 2023 Jan;66(1):241-246. doi: 10.1007/s00125-022-05805-3. Epub 2022 Oct 4. PMID 36194251
- [Derived] Neuman V, Cinek O, Funda DP, Hudcovic T, Golias J, Kramna L, Petruzelkova L, Pruhova S, Sumnik Z. Human gut microbiota transferred to germ-free NOD mice modulate the progression towards type 1 diabetes regardless of the pace of beta cell function loss in the donor. Diabetologia. 2019 Jul;62(7):1291-1296. doi: 10.1007/s00125-019-4869-2. Epub 2019 Apr 25. PMID 31025045

RESULTS

PARTICIPANT FLOW:
Groups:
- Gluten-free Diet: Gluten-free diet for pediatric patients with type 1 diabetes
- Conventional Diet: Conventional gluten-containing diet for pediatric patients with type 1 diabetes
Period: Overall Study
Arm/Group | Gluten-free Diet | Conventional Diet
Started | 26 | 19
Completed | 20 | 19
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gluten-free Diet | Conventional Diet | Total
Number analyzed (Participants) | 26 | 19 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 19 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (3.2) | 10.1 (3.5) | 10.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 26 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in C-peptide Area Under the Curve Measured by Mixed-meal Tolerance Test (MMTT) Between Group on GFD and Standard Gluten-containing Diet.
Description: Area under the curve of C-peptide in MMT test at 0, 30, 60, 90 and 120 minutes.
Time Frame: Month 1 (baseline) - Month 12 (end of intervention)
Measure: Mean (Standard Deviation); unit: pmol*min/l
Arm/Group | Gluten-free Diet | Conventional Diet
Number analyzed (Participants) | 20 | 19
pmol*min/l | 1539 (1255) | 1173 (1006)
Statistical Analysis 1: Comparison: Gluten-free Diet vs Conventional Diet; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 205, 95% CI 2-sided [-223 to 633]

2. Secondary Outcome: Changes in Mean HbA1c at 6 and 12 Months Relative to Baseline at Month 1.
Time Frame: Month 1 (baseline) - Month 6 - Month 12 (end of intervention)
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Gluten-free Diet | Conventional Diet
Number analyzed (Participants) | 20 | 19
mmol/mol
  HbA1c at 6 months | 44.8 (6.3) | 47.2 (8.3)
  HbA1c at 12 months | 44 (9.5) | 52.2 (10.6)
Statistical Analysis 1: Comparison: Gluten-free Diet vs Conventional Diet; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -7.8, 95% CI 2-sided [-14.1 to -1.6]

3. Secondary Outcome: Changes in Mean Insulin Dose at 6 and 12 Months Relative to Baseline at Month 1.
Time Frame: Month 1 (baseline) - Month 6 - Month 12 (end of intervention)
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Gluten-free Diet | Conventional Diet
Number analyzed (Participants) | 20 | 19
U/kg/day
  Insulin dose at 6 months | 0.41 (0.17) | 0.62 (0.23)
  Insulin dose at 12 months | 0.50 (0.22) | 0.75 (0.34)
Statistical Analysis 1: Comparison: Gluten-free Diet vs Conventional Diet; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.31 to 0.01]

4. Secondary Outcome: Changes in Immunological Parameters (FoxP3 Tregs, Th1 and Th17 Counts) at 12 Months Relative to Baseline at Month 1.
Time Frame: Month 1 (baseline) - Month 12 (end of intervention)
Measure: Mean (Standard Deviation); unit: % of cells
Arm/Group | Gluten-free Diet | Conventional Diet
Number analyzed (Participants) | 20 | 19
% of cells
  TEMRA cells at 12 months | 8 (2.2) | 12.5 (3.5)
  T-regulatory cells type 1 at 12 months | 1.02 (0.63) | 0.46 (0.16)
Statistical Analysis 1: Comparison: Gluten-free Diet vs Conventional Diet; Test type: Superiority; p < 0.05, t-test, 1 sided

5. Secondary Outcome: Differences in Fecal Microbiome Between Children on Normal Diet and Children on Gluten-free Diet Over the First Year of Diabetes Duration
Description: Measures are shown as pooled values at all timepoints during the intervention period compared to control group throughout the same time-period.
Time Frame: Month 1 (before intervention) - Pooled values throughout the intervention (months 3-12) - Month 15 (after intervention)
Measure: Number; unit: Percentage of microbes
Arm/Group | Gluten-free Diet | Conventional Diet
Number analyzed (Participants) | 22 | 19
Percentage of microbes
  Bifidobacterium | 3.3 | 8
  Roseburia | 3.2 | 1.2
  Lachnospira | 1.01 | 0.21
Statistical Analysis 1: Comparison: Gluten-free Diet vs Conventional Diet; Test type: Superiority; p < 0.05, ANOVA — After Benjamini-Hochberg correction for multiple comparisons

ADVERSE EVENTS:
Time Frame: 15 months
Description: Specific AE questionnaire given at each visit (i.e. in 3 months periods).
Arm/Group | Gluten-free Diet | Conventional Diet
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/19
Other Adverse Events (participants affected / at risk) | 0/26 | 0/19

LIMITATIONS AND CAVEATS:
The main limitation is the lack of randomization. Second, the study did not achieve the sample size needed for sufficient power according to the pre-study power analysis. Furthermore, the duration of the study might have been too short for the assessment of the long-term effect of the GFD on the course of T1D.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT02867436/Prot_SAP_000.pdf